CLINICAL TRIAL: NCT03127046
Title: A Randomized, Open-label, Single Dose, 3-way Crossover Study to Evaluate the Drug-drug Interaction Between Aceclofenac 200 mg and Esomeprazole 20 mg in Healthy Male Volunteers
Brief Title: Drug-drug Interaction Between Aceclofenac 200 mg and Esomeprazole 20 mg in Healthy Male Volunteers
Acronym: DW6008
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW6008-I-1
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — aceclofenac; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1 (Experimental): Aceclofenac → Esomeprazole → Concomitant of Aceclofenac and esomeprazole
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole
- Group 2 (Experimental): Concomitant of Aceclofenac and esomeprazole→Aceclofenac→ Esomeprazole
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole
- Group 3 (Experimental): Esomeprazole →Concomitant of Aceclofenac and esomeprazole→ Aceclofenac
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole
- Group 4 (Experimental): Concomitant of Aceclofenac and esomeprazole→Esomeprazole→Aceclofenac
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole
- Group 5 (Experimental): Esomeprazole→Aceclofenac→ Concomitant of Aceclofenac and esomeprazole
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole
- Group 6 (Experimental): Aceclofenac→Concomitant of Aceclofenac and esomeprazole→Esomeprazole
  Interventions: Drug: Aceclofenac; Drug: Esomeprazole; Drug: Aceclofenac and Esomeprazole

INTERVENTIONS:
Drug: Aceclofenac — Oral single dose administration of aceclofenac 200mg
  Other Names: Airtal tablet
Drug: Esomeprazole — Oral single dose administration of aceclofenac 200mg
  Other Names: Nexium tablet
Drug: Aceclofenac and Esomeprazole — Oral single dose administration of aceclofenac 200mg and esomeprazole concomitant
  Other Names: Airtal and Nexium concomitant

SUMMARY:
To evaluate the drug-drug interaction between aceclofena and esomeprazole

DETAILED DESCRIPTION:
A randomized, open-label, single dose, 3-way crossover study to evaluate the drug-drug interaction between Aceclofenac 200 mg and Esomeprazole 20 mg in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* A healthy man over 19 years old
* Body Mass Index(BMI)=17.5~30.5kg/m2, one with weight of more than 55kg (BMI= kg/(m)2)
* Congenital or chronic diseases within the last three years, there is no medical examination results of popular characters with no psychotic symptoms or findings
* Depending on the nature of the drug your doctor check conducted hematology, blood chemistry, urinalysis and laboratory tests, including an electrocardiogram(EKG) performed during screening tests such as a suitable test subjects who judged
* The purpose of the test participants prior to testing, information, and to hear about the free will fully explain to participate in this study, according to the Institutional Review Board(IRB)-approved consent form signed by the parties in writing

Exclusion Criteria:

* one with clinically significant blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic disease (but ,except for untreated seasonal allergies of asymptomatic at the time of administration) with medical history or evidence
* one with gastrointestinal disease(Such as esophageal stricture or achalasia of the esophagus disease, Crohn disease) to affect drug absorption or surgery(but, excluding simple appendectomy or hernia surgery) with medical history
* Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 2 times the upper limit of the normal range
* Within 6 months, 210 g / week of alcohol in excess of a history of regular characters (beer (5%) 1 cup (250 mL) = 10 g, soju(20%) 1 cup (50 mL) = 8 g, Wine (12%) 1 cup (125 mL) = 12 g)
* Take part in other clinical trials within three months
* Systolic Blood Pressure(SBP) ≥ 140 mmHg or Diastolic Blood Pressure (DBP) ≥ 90 mmHg
* The great history of alcohol or drug abuse within 1 year
* Taking medication of drug-metabolizing enzymes that are known to significantly induce or inhibit within 30 days
* More than 20 cigarettes a day smoker
* Taking medication of a prescription drug or nonprescription within 10 days,
* Within two months the whole blood donation have, within one month of the apheresis donation have
* Participate in clinical trials to test drug administration and may be at increased risk due to interpretation of test results, or may interfere with severe supply / chronic medical or mental condition or abnormal laboratory test values in character

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-04-23 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 24hours
  Maximum concentration of aceclofenac and esomeprazole in plasma
AUClast | up to 24hours
  Area under the plasma concentration versus time curve to last time of aceclofenac and esomeprazole in plasma

SECONDARY OUTCOMES:
t1/2 | up to 24hours
  Terminal half-time of aceclofenac and esomeprazole in plasma
Tmax | up to 24hours
  Time to reach Cmax of aceclofenac and esomeprazole in plasma
CL/F | up to 24hours
  Apparent clearance of aceclofenac and esomeprazole
Vd/F | up to 24hours
  Apparent volume of distribution of aceclofenac and esomeprazole

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, PhD, Principal Investigator — Chonbuk National University Hospital in Korea
Locations (1):
- Chonbuk National University Hospital., Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No